CLINICAL TRIAL: NCT06153654
Title: Role of the Nasal Microbiota in Obesity - the microNASA Study
Brief Title: Role of the Nasal Environment in Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Katharina Timper (Other)
Responsible Party: Sponsor-Investigator, Katharina Timper, Prof. Dr. med., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 2021-01090
Record Dates: First submitted 2022-01-28; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Adiposity
Keywords: Adiposity; Olfactory Function; Microbiome
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese: Obese participants with BMI >30
- Lean: Lean participants with a BMI <25
- Bariatric: Participants with scheduled bariatric surgery.

SUMMARY:
The primary aim of this study is to investigate the nasal environment in obese and lean individuals.

ELIGIBILITY:
Inclusion Criteria:

N=50 adult male and female patients with obesity will be included in this study.

Inclusion criteria:

Inclusion criteria:

* Age 18-55 years
* Written informed consent
* BMI > 30 kg/m2

N=50 adult lean patients age- and sex-matched to the group of obese patients will be included in this study.

Inclusion criteria:

* Age 18-55 years
* Written informed consent
* BMI 18-25 kg/m2

N=50 adult male and female patients with obesity with scheduled bariatric will be included in this study

Inclusion criteria:

* Age 18-55 years
* Written informed consent
* BMI > 35 kg/m2

Exclusion Criteria:

* Smoking
* Chronic or acute sinusitis
* Surgical intervention of the nasal cavity or the paranasal sinus
* Use of antibiotics within the last 31 days18
* Current illicit drug abuse including daily marijuana or CBD consumption (≤ 24 g of alcohol per day allowed)
* Any kind of severe chronic disease (e.g. severe heart failure, active cancer disease)
* Use of any kind of decongestant more than twice a week
* Use of cortisone-containing nasal spray within the last 3 months
* Acute allergic rhinitis
* History of neurodegenerative diseases
* History of severe head trauma
* Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2)

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Male and female participants between the age of 18-55. 50 participants with obesity, 50 lean participants (age- and sex-matched), 50 patients with schedueled bariatric surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Difference in nasal microbiota composition | 6 Months
  The microbiome of the nasal cavity will be analyzed by isolating DNA from Nasal Swabs through amplicon sequencing. We will define the primary endpoint as the difference in nasal microbiome in obese vs. sex- and age-matched lean control individuals.

SECONDARY OUTCOMES:
Change in nasal microbiota Composition after bariatric surgery | 24 Months
  The microbiome of the nasal cavity will be analyzed by isolating DNA from Nasal Swabs through amplicon sequencing. We will define the primary endpoint as changes in nasal microbiome in obese patients before and 1, 3, 6 and 12 month after bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Timper, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland